CLINICAL TRIAL: NCT05594381
Title: A Prospective, Open-label, Single-Arm, Phase II Study on Biomarkers for Predicting the Efficacy of Neoadjuvant Sintilimab in Combination With Tegafur and Oxaliplatin (SOX) for cStage III Gastric or Gastroesophageal Junction Adenocarcinoma.
Brief Title: A Biomarker Study for Predicting the Efficacy of Neoadjuvant Sintilimab Plus SOX for Gastric Adenocarcinoma.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Innovent Biologics (Suzhou) Co. Ltd. (Industry); Nanjing Geneseeq Technology Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: JSGCLB-2201
Record Dates: First submitted 2022-09-29; First posted 2022-10-26 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Gastric Cancer
Keywords: Gastric Cancer with cStage III; Circulating tumor DNA; Neoadjuvant immunotherapy plus chemotherapy; Evaluation biomarkers
MeSH Terms: conditions — Stomach Neoplasms | interventions — sintilimab; Oxaliplatin; Tegafur

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant Sintilimab plus SOX therapy (Experimental): All enrolled subjects were treated with Sintilimab combined with SOX regimen (Oxaliplatin plus Tegafur) for 3 cycles and then underwent radical surgery.
  Peripheral blood from all patients will be collected at the following 5 time points: before neoadjuvant therapy (within 3 days before the first dose); before the start of the third cycle of neoadjuvant therapy (within 3 days); before surgery (within 7 days) and after surgery (within 3-7 days). Plasma was tested for ctDNA. All subjects were further stratified according to the detection results of ctDNA and their changes during the neoadjuvant treatment period.
  After operation, sintilimab combined with SOX therapy was continued for 5 cycles according to the original plan (if the preoperative treatment did not reach 3 cycles, it should be supplemented to 8 cycles)
  Interventions: Drug: Sintilimab

INTERVENTIONS:
Drug: Sintilimab — Neoadjuvant treatment method: Sintilimab 200 mg, i.v., d1 + oxaliplatin 130 mg/m2, d1, i.v., + Tegafur 40 mg po, bid, d1-14; 3-week course; Neoadjuvant therapy: 3 courses of preoperative SOX chemotherapy (oxaliplatin+Tegafur) + PD-1 monoclonal antibody (Sintilimab).
  After the 2nd and 3rd cycles of neoadjuvant therapy (6-9 weeks from the start of treatment), imaging effects and feasibility of radical surgery were performed respectively; The operation time is arranged within 2-6 weeks after the last administration of neoadjuvant therapy, and the operation method is selected by the surgeon according to the actual needs; The postoperative treatment plan is the same as the preoperative neoadjuvant treatment plan, and the SOX+Sintilimab will continue to be given until the full 8 cycles (including the preoperative 3 cycles).
  Other Names: Oxaliplatin; Tegafur; Radical gastrectomy with D2 lymph node dissection

SUMMARY:
Recently, a number of clinical studies were carried out to evaluate the therapeutic effects of PD-1 antibodies combined with chemotherapy as preoperative neoadjuvant therapy of gastric cancer (GC) worldwide. Indicators such as PD-L1 expression, TMB and MSI are currently used to evaluate the efficacy of PD-1/PD-L1 monoclonal antibody therapy. However, these biomarkers are mainly used in patients with metastatic and unresectable tumors, and the conclusions obtained in different studies are still partially contradictory, failing to accurately guide the treatment. Therefore, it is urgent to explore highly sensitive and specific biomarkers that can be used to monitor the efficacy of neoadjuvant immunotherapy for GC.The present clinical trial aims to use ctDNA dynamic monitoring combined with multi-omics methods to evaluate PD-1 monoclonal antibody (sintilimab) combined with SOX neoadjuvant therapy for clinical stage III gastric/gastroesophageal junction adenocarcinoma. In order to identify the suitable population for neoadjuvant immunotherapy for locally advanced and resectable G/GEJ adenocarcinoma.

DETAILED DESCRIPTION:
At present, radical surgery is still the only way to cure Gastric Cancer（GC）, but the surgical resection rate is low, and the R0 resection rate is about 70-80%. The postoperative recurrence rate of patients with stage II and above is high. To improve the surgical resection rate, seek more effective treatment. The other treatment therapeutics are the direction of development of GC treatment research. Neoadjuvant therapy for GC can reduce tumor stage and increase the likelihood of complete tumor resection to achieve maximum pathological response. Neoadjuvant chemotherapy followed with surgery has been written into the NCCN guidelines for GC. Since China, the United States and Japan successively approved PD-1 monoclonal antibody for the treatment of unresectable and/or metastatic GC and gastroesophageal junction adenocarcinoma (G/GEJ adenocarcinoma), a number of clinical studies about the therapeutic effects of PD-1 antibodies combined with chemotherapy as preoperative neoadjuvant therapy are carring out worldwide. A single-arm phase II clinical study has demonstrated that the Sintilimab,which is the only one PD-1 mAb that has the indication for first-line treatment of GC in China, combined with oxaliplatin and capecitabine in neoadjuvant treatment of locally advance resectable GC. The treatment showed encouraging pCR rates and a good safety profile. However, how to select suitable patients for neoadjuvant immunotherapy is the focus of current research.

Indicators such as PD-L1 expression, tumor mutation burden, and microsatellite stability are currently considered to be the average indicators of the efficacy of PD-1/PD-L1 monoclonal antibody therapy. However, according to the NCCN guidelines, these biomarkers are mainly used in patients with advanced postoperative tumors, and the conclusions obtained in different studies such as KEYNOTE-061 and KEYNOTE-062 are still partially contradictory, failing to accurately guide the treatment. Therefore, it is urgent to explore highly sensitive and specific indicators that can be used to monitor the efficacy of neoadjuvant immunotherapy for GC.

This study intends to dynamically detect gene mutations, protein expressions and tumor images in G/GEJ tumor tissues and blood samples before, under and after neoadjuvant therapy by using ctDNA targeted sequencing combined with multi-omics technology. Through independent and association analysis and building risk models, biomarkers with significant predictive effects on the curative effect of neoadjuvant immunotherapy were found, so as to identify the suitable population for neoadjuvant immunotherapy for locally advanced and resectable G/GEJ adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. G/GEJ adenocarcinoma patients aged 18-75 years old, male or female;
2. Patients with cStage III by abdominal CT and intraoperative assessment, and G/GEJ adenocarcinoma diagnosed by gastroscope and pathology (regardless of HER-2 expression), and gastroesophageal junction (GEJ) cancer only allows Siewert III Type II, and Siewert type II subjects who did not require combined thoracotomy were enrolled.
3. Before enrollment, a gastrointestinal surgeon and an imaging technologist will jointly evaluate the tumor as cStage III and be eligible for R0 resection for the purpose of cure;
4. The initial diagnosis has not been treated;
5. Expected survival period ≥ 3 months;
6. According to the RECIST v1.1 criteria (see Annex 3 for details), there are measurable tumor lesions;
7. The ECOG PS score within 7 days of the first medication (see Annex 4 for details) is 0-1;
8. The heart function is good, and resection for curative purpose can be performed. Patients with underlying ischemic, valvular, or other serious cardiac disease should be evaluated preoperatively by a cardiologist if clinically indicated;
9. Those who have used anti-tumor traditional Chinese medicines, proprietary Chinese medicines, and immunomodulators (such as thymosin, lentinan, interleukin-12, etc.) must be ≥ 2 weeks away from the start of the study medication.
10. To have sufficient organ function, subjects must meet the following laboratory indicators:1) The absolute value of neutrophils (ANC) is ≥1.5x109/L without the use of granulocyte colony-stimulating factor in the past 14 days; 2) Platelets ≥100×109/L without blood transfusion in the past 14 days; 3) Hemoglobin>9g/dL without blood transfusion or use of erythropoietin in the past 14 days; 4) Total bilirubin≤1.5×ULN; if total bilirubin>1.5×ULN but direct bilirubin≤ULN, it is also allowed to enter the group; 5) Aspartate aminotransferase (AST), alanine aminotransferase (ALT) in ≤2.5×ULN; 6) Serum creatinine ≤1.5×ULN and creatinine clearance rate (calculated by Cockcroft-Gault formula) ≥60 ml/min; 7) Good coagulation function, defined as international normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 times ULN; 8) Normal thyroid function, defined as Thyroid Stimulating Hormone (TSH) within the normal range. If the baseline TSH exceeds the normal range, subjects with total T3 (or FT3) and FT4 within the normal range can also be enrolled; 9) Myocardial enzyme spectrum is within the normal range (if the investigator comprehensively judges that the simple laboratory abnormality does not have clinical significance, it is also allowed to enter the group);
11. Thyroid function indicators: Thyroid-stimulating hormone (TSH), free thyroxine (FT3/FT4) in the normal range or mild and no clinically significant abnormalities;
12. Weight above 40 kg (including 40 kg), or BMI>18.5;
13. Female patients must meet:

    * Menopausal (defined as the absence of menstruation for at least 1 year and no other confirmed cause other than menopause) status, or who have undergone surgical sterilization (removal of ovaries and/or uterus), or are fertile patients must meet both of the following requirements:
    * Serum pregnancy test results must be negative within 7 days prior to the first dose;
    * Consent to use contraception with an annual failure rate of < 1% or maintain abstinence (avoid heterosexual intercourse) (from signing the informed consent form to at least 120 days after the last dose of the trial drug, and at least 6 months after surgery (annual failure rate < 1%) Contraceptive methods include bilateral tubal ligation, male sterilization, proper use of hormonal contraceptives that inhibit ovulation, hormone-releasing IUDs, and copper-containing IUDs.);
    * Do not breastfeed.
14. Male patients must meet:

    Consent to abstinence (avoid heterosexual intercourse) or use contraceptive measures as follows: When the partner is a female of childbearing age or the partner is pregnant, the male patient must remain abstinent for at least 120 days after the last dose of the trial drug and for at least 120 days after surgery or Use condoms correctly. The reliability of sexual abstinence should be evaluated with reference to the duration of clinical studies, patient preferences, and lifestyle. Periodic abstinence (e.g., calendar days, ovulation, basal body temperature, or post-ovulatory contraceptive methods) and ejaculation are inappropriate contraceptive methods;
15. The subjects read and fully understand the patient instructions and signed the informed consent.

Exclusion Criteria:

1. The patient has other malignant tumors in the past (within 5 years) or at the same time. Cured localized tumors, such as basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, carcinoma in situ of the prostate, carcinoma in situ of the cervix, carcinoma in situ of the breast, stage I lung cancer, stage I colorectal cancer, etc. ;
2. Patients who are going to undergo or have received organ or bone marrow transplantation in the past;
3. Have undergone blood transfusion within 2 weeks before the first drug, or have a history of bleeding, and have any bleeding event with a severe grade of CTCAE4.0 grade 3 or above within 4 weeks before screening;
4. Patients with abnormal coagulation function and bleeding tendency (INR is >1.5 in the absence of anticoagulants); patients treated with anticoagulants or vitamin K antagonists such as warfarin, heparin or their analogs ; On the premise of prothrombin time international normalized ratio (INR) ≤ 1.5, low-dose warfarin (1 mg orally, once a day) or low-dose aspirin (no more than 100 mg per day) is allowed for prophylaxis. ;
5. Arterial/venous thrombosis events occurred within 6 months before screening, such as cerebrovascular accident (including temporary ischemic attack), deep vein thrombosis (venous thrombosis caused by venous intubation due to previous chemotherapy and has been cured by the investigator's judgment excluding those) and pulmonary embolism, etc.;
6. Myocardial infarction and poorly controlled arrhythmia (including QTc interval ≥ 450 ms for men and ≥ 470 ms for women) within 6 months before the first medication (QTc interval is calculated by Fridericia formula);
7. The presence of NYHA standard III to IV cardiac insufficiency or cardiac ultrasound examination: LVEF (left ventricular ejection fraction) <50%;
8. Urine routine indicates urine protein ≥++ and confirmed 24-hour urine protein quantification >1.0 g;
9. There are multiple factors that affect oral drugs (such as inability to swallow, chronic diarrhea and intestinal obstruction, etc.);
10. Pleural effusion or ascites with clinical symptoms requiring clinical intervention;
11. Human immunodeficiency virus (HIV) infection;
12. Suffering from active pulmonary tuberculosis;
13. Long-term unhealed wounds or incompletely healed fractures;
14. Patients with past and current interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, severely impaired lung function, etc., which may interfere with the detection and treatment of suspected drug-related pulmonary toxicity;
15. There is a known active or suspected autoimmune disease, except those who are in a stable state of the disease at the time of enrollment (systemic immunosuppressive therapy is not required);
16. History of severe chronic autoimmune diseases, such as systemic lupus erythematosus; history of ulcerative colitis, Crohn's disease and other inflammatory bowel diseases; history of chronic diarrheal diseases such as irritable bowel syndrome; History of sarcoidosis or tuberculosis; active hepatitis B, hepatitis C and HIV infection; well-controlled non-serious immune diseases, such as dermatitis, arthritis, psoriasis, etc. can be enrolled. Hepatitis B virus titer < 500copy/ml can be enrolled;
17. Patients who need to receive systemic corticosteroids (> 10 mg/day efficacy dose of prednisone) or other immunosuppressive drugs within 14 days before the first dose or during the study. However, the following conditions are allowed: in the absence of active autoimmune disease, patients are allowed to use topical or inhaled steroids, or adrenal hormone replacement therapy at a dose of ≤ 10 mg/day of prednisone efficacy;
18. Any active infection that requires systemic anti-infective treatment within 14 days before the first dose; except for prophylactic antibiotic treatment (such as the prevention of urinary tract infection or chronic obstructive pulmonary disease);
19. Received treatment with live vaccines within 28 days before the first dose; except for inactivated viral vaccines for seasonal influenza;
20. Received other antibody/drug therapy targeting immune checkpoints in the past, such as PD-1, PD-L1, CTLA4, etc.;
21. Are receiving other clinical research treatments, or planning to start the treatment in this study less than 1 month after the end of the treatment in the previous clinical study;
22. Known history of severe allergy to any monoclonal antibody or study drug excipients;
23. The patient has a history of alcoholism, drug use and drug abuse. Patients who have stopped drinking alcohol can be enrolled;
24. Patients who do not follow doctor's orders, do not take medicines as prescribed, or have incomplete information, which may affect the judgment of efficacy or safety;
25. Pregnant or lactating female patients;
26. There are patients who may increase the risk of participating in research and research medication, or have other severe, acute and chronic diseases, who are judged by the investigator and are not suitable for participating in clinical research.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate (pCR) | an average of 6 months.
  pCR rate is the proportion of patients who have no residual viable tumor in the resected specimens.
  The primary aim of the study is to test the hypothesis that after neoadjuvant therapy，patients with ctDNA clearance result in a higher rate of pCR.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | an average of 4 months.
  ORR refers to the proportion of subjects with confirmed best overall response of complete response (CR) or partial response (PR), based on RECIST 1.1 DCR refers to the percentage of confirmed complete remission (CR), partial remission (PR), and stable disease (SD) cases among patients with evaluable response.
Disease Control Rate (DCR) | an average of 4 months.
  DCR refers to the proportion (%) of patients with at least one visit response of complete response (CR) or partial response (PR), or stable disease (SD) based on RECIST1.1
Major pathological response rate (MPR) | after surgery，an average of 6 months.
  MPR refers to as the proportion of patients with less than 10% viable tumour at resection.
Tumor Regression Grade (TRG) | an average of 6 months.
  TGR grading using the Becker criteria as follows: TRG1a (no residual tumor), equivalent to pCR; TRG1b (<10% residual tumor); TRG2 (10%-50% residual tumor); TRG3 (>50% residual tumor).
R0 resection rate | an average of 6 months.
  R0 resection rate refers to the proportion of all patients with negative margins under the microscope of tumor specimens after surgery to the total number of participants.
T(tumor) and/or N(node) downstaging rate | an average of 6 months.
  T(tumor) and/or N(node) downstaging is defined as the postoperative pathological T and/or N stage lower than the original stage by imaging before neoadjuvant treatment.
30-day post-operative surgical complication rate | 30 days postoperation.
  based on the Clavien-Dindo classification
Disease-free survival (DFS) | up to 2 years after surgery.
  Disease-free survival was defined as from the start of surgery to disease recurrence or death (for any reason).
Overall Survival（OS） | up to 2 years after surgery.
  Overall survival was defined as the date from patient enrollment to death of any cause.
Incidence of Treatment-Emergent Adverse Events（Safety） | up to 2 years after surgery.
  Safety as measured by number and grade of adverse events. Numbers of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs), events will be classified according to CTCAE V5.0.

OTHER OUTCOMES:
Relationship between the numerical changes of ctDNA during neoadjuvant immunotherapy plus chemotherapy and postoperative pathological remission rate | an average of 6 months.
  To evaluate whether the trend of changes in ctDNA values during neoadjuvant immunotherapy combined with chemotherapy can be used to predict postoperative pathological response rate.
Genomic changes of ctDNA | an average of 6 months.
  To dynamically evaluate the ctDNA profiles by next-generation sequencing and illustrate the genomic changes of ctDNA at baseline, during and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Zekuan Xu, PhD, Study Chair — The First Affiliated Hospital with Nanjing Medical University

IPD SHARING:
Plan to Share IPD: No